CLINICAL TRIAL: NCT04591327
Title: Determination of the Effects of General Anesthesia and Spinal Anesthesia Applied in Elective Cesarean Operations on Postoperative Atelectasis by Lung Ultrasonography
Brief Title: Atelectasis by Lung Ultrasonography in Cesarean Sections
Status: Completed | Type: Observational
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ERHAN KARACA, Principal Investigator, Derince Training and Research Hospital
Other Study IDs: U1111-1258-9377
Record Dates: First submitted 2020-10-04; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Atelectasis; Cesarean Section
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- general anesthesia
  Interventions: Procedure: The Effect of General Anesthesia and Spinal Anesthesia on Postoperative Atelectasis by Lung Ultrasonography in Cesarean Sections
- spinal anesthesia
  Interventions: Procedure: The Effect of General Anesthesia and Spinal Anesthesia on Postoperative Atelectasis by Lung Ultrasonography in Cesarean Sections

INTERVENTIONS:
Procedure: The Effect of General Anesthesia and Spinal Anesthesia on Postoperative Atelectasis by Lung Ultrasonography in Cesarean Sections — Preoperative lung ultrasound will be performed on all patients and baseline values will be recorded. The sensory block level under T10 of the patients who underwent spinal anesthesia in the postoperative period lung ultrasonography will be done after regression. In the postoperative period, lung ultrasonography will be performed in patients undergoing spinal anesthesia when the sensory block level is below T10. In the general anesthesia group, when the neuromuscular block is completely reversed and the Aldrete score is> 9, lung ultrasonography will be performed. The degree of atelectasis will be determined according to the modified LUS score.

SUMMARY:
In this study aimed to demonstrate that atelectasis developing in the perioperative period of patients undergoing elective cesarean surgery with spinal or general anesthesia methods using lung ultrasound. After Preoperative lung ultrasounds of patients is done, the cesarean operation will be completed with spinal or general anesthesia. In the postoperative period, control lung ultrasounds will be performed and the ultrasound results will be compared in terms of atelectasis in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-40 years
* 37-40 weeks pregnant
* ASA II because of pregnancy

Exclusion Criteria:

* Emergency cesarean sections
* who refuse to participate in the study
* with chronic disease
* Smoker
* with chest deformity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Between 18-40 years old, 37-40 weeks pregnant, ASA II because of pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
incidence of the postoperative atelectasis | two months

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Derince Train and Research Hospital, Kocaeli, Turkey (Türkiye)